CLINICAL TRIAL: NCT05088889
Title: Maintenance Ipilimumab + Nivolumab Post Induction Chemotherapy + SBRT for First Line
Brief Title: Maintenance Ipilimumab + Nivolumab Post Induction Chemotherapy + SBRT for First Line Treatment Stage IV Pancreatic Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Dr. Talia Golan, Medical diractor of phase 1 clinical trials unit and Sheba pancreatic cancer program, The Chaim Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA184-604
Record Dates: First submitted 2021-06-22; First posted 2021-10-22 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Stage IV Pancreatic Cancer
Keywords: Pancreatic adenocarcinoma; SBRT (Stereotactic body radiation therapy); immunotherapy; RECIST1.1 (Response Evaluation Criteria in Solid Tumours V1.1)
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Nivolumab; Ipilimumab; Radiosurgery; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study arm (Experimental): Study treatments include SBRT (Stereotactic radiation therapy) to one primary/metastatic tumor (3 fractions of 8Gy) , and ipilimumab (1mg/kg every six weeks) + nivolumab (360mg every three weeks) .
  Every 8 weeks patients will be assessed for response; responders will continue ipilimumab + nivolumab until disease progression, non-responders will receive very low dose radiation (2Gy single fraction to metastatic lesions of choice) prior to continuing ipilimumab + nivolumab .
  Interventions: Drug: Nivolumab; Drug: ipilimumab; Radiation: Stereotactic body radiation therapy; Radiation: Low dose irradiation

INTERVENTIONS:
Drug: Nivolumab — Nivolumab administered IV over 30 minutes at a dose of 360mg every 3 weeks
Drug: ipilimumab — Ipilimumab administered IV over 30 minutes at 1 mg/kg every 6 weeks
Radiation: Stereotactic body radiation therapy — Three fractions of 8 Gy, treated on alternate days
  Other Names: SBRT
Radiation: Low dose irradiation — a single fraction of 2Gy will be given to the metastatic lesions at first progression

SUMMARY:
In this study we aim to test the efficacy of a combined and novel approach including induction chemotherapy (per standard of care) followed by SBRT and maintenance ipililumab + nivolumab in the first line setting of stage IV PDAC.

Study Hypothesis:

Cytotoxic chemotherapy followed by hypofractionated radiotherapy will sensitize pancreatic cancer to immunotherapy consisting of combined PD-1 and CTLA4 blockade. We hypothesize that direct targeting of the pancreatic cancer cells by chemotherapy and hypofractionated radiotherapy is necessary for initial anti-tumor response. Furthermore, the combination of immunotherapy as a maintenance strategy will have profound anti-tumor efficacy in this setting.

Implications of hypothesis:

* Improved response rate above historical controls
* Lengthened progression-free survival
* Improved overall-survival

Exploratory Hypothesis:

We hypothesize that baseline markers of immune activation such as Tumor Infiltrating Lymphocytes and CD8+ lymphocytes will correlate with response to ipililumab + nivolumab and that responders will have distinct tumor immune phenotype as determined by immunohistochemistry and gene expression profiling compared to nonresponders.

DETAILED DESCRIPTION:
This is a single arm, single institution study, which aims to evaluate the efficacy and safety of combination therapy with radiosurgery nivolumab and ipilimumab as a maintenance regimen following first line induction chemotherapy in patients with metastatic pancreatic cancer.

Chemotherapy will be administrated for a minimum of 4 cycles. Patients who have not progressed on chemotherapy will receive SBRT to one primary/metastatic tumor, followed by ipilimumab (1mg/kg every six weeks) + nivolumab (360mg every three weeks). After a further 8 weeks patients will be assessed for response; responders will continue ipilimumab + nivolumab until disease progression, non-responders will receive very low dose radiation to metastatic sites (this will only be allowed once) prior to continuing ipilimumab + nivolumab until disease progression. Immunotherapy will be continued until disease progression or up to 24 months in the absence of disease progression or unacceptable toxicity.

Study rationale Overall rational in Brief Although there is evidence for that the immune system plays an active role in pancreatic cancer, until now checkpoint inhibitors have yet to demonstrate efficacy in this population. We hypothesize that combining irradiation along with checkpoint inhibition in a patient population demonstrating stable disease in a first line setting will be a novel approach towards the treatment of pancreatic cancer.

Rationale for Combining Nivolumab and Ipilimumab The roles of CTLA-4 and PD-1 in inhibiting antitumor responses are largely distinct. Whereas CTLA-4 is thought to regulate T-cell proliferation early in the immune response, primarily in lymph nodes, PD-1 suppresses T cells at a later stage in the immune response, primarily in peripheral tissues.

Preclinical data indicate that the combination of PD-1 and CTLA-4 receptor blockade may improve antitumor activity.

Encouraging response rates for the combination of nivolumab and ipilimumab have been demonstrated in several types of cancer such as melanoma, renal cell carcinoma, and non-small cell lung cancer.

Due to toxicity concerns regarding the combination of nivolumab and ipilimumab, several different doses and schedules were evaluated in a phase 1 study as first-line therapy in patients with advanced NSCLC (CA209012). This study identified an alternative schedule with an acceptable tolerability profile (28% grade 3-4 toxicity) and encouraging activity (31% overall response rate) - nivolumab 360 mg/kg every 3 weeks plus ipilimumab 1 mg/kg every 6 weeks, and has therefore been adopted in this protocol.

Rationale for Combining Radiosurgery with anti-PD-1 and anti-CTLA-4 High-dose radiation (such as used in stereotactic radiation body therapy - SBRT) induces DNA damage and cell death. Radiation alone appears to induce a systemic immune response.

The biologic rationale behind the strategy is that radiation will cause release of immunogenic tumor-antigens from dying tumor cells, which will be processed by cells of the adaptive immune system, eventually promoting tumor-specific targeting of the tumor by the immune system. Success of this strategy will hopefully induce and augment the rarely seen abscopal effect. One possible explanation is that radiation alone rarely induces a rich immune infiltrate into the dying tumor.

Radiation dose and fractionation schedules for optimal synergy between radiotherapy and immunotherapy are not well defined. Three fractions of 8 Gy has been successfully combined with anti-CTLA-4 therapy in mice, and has emerged as a popular regimen for radiation - immunotherapy trials, and has therefore been adopted in this protocol.

Study Population Estimated accrual - 10 patients. The patients for the study will be identified from the pancreatic cancer clinics at Sheba Medical Center with advanced pancreatic cancer (stage IV) in the first-line setting.

Approximately 17 patients will be initially evaluated in the first line setting. We estimate that approximately 50-60% will not progress at three months and they will continue to receive the study treatment. Only the non-progressors who receive SBRT and combination immunotherapy will be evaluated in the ITT population.

TREATMENT PLAN:

Stereotactic radiosurgery Simulation will be performed in accordance with the target lesion location, with 3D or 4D CT as appropriate. Three fractions of 8 Gy, treated on alternate days (in exceptional circumstances, may treat on consecutive days).

Nivolumab and Ipilimumab Nivolumab administered IV over 30 minutes at a dose of 360mg every 3 weeks. Ipilimumab administered IV over 30 minutes at 1 mg/kg every 6 weeks following the administration of nivolumab. On the day of infusion, nivolumab is to be administered first. Ipilimumab will start at least 30 minutes after completion of the nivolumab infusion. Nivolumab and ipilimumab will be continued until the progression of disease, discontinuation due to toxicity, withdrawal of consent, or study closure. In any event medication will not be continued beyond 24 months. Subjects may discontinue only ipilimumab and continue treatment with nivolumab if certain circumstances are met. Treatment beyond initial investigator assessed RECIST v1.1 defined progression 2 is permitted if the subject has investigator assessed clinical benefit and is tolerating nivolumab and ipilimumab.

Low dose irradiation at first progression At time of 1st progression, at physician's discretion, a single fraction of low dose irradiation (2Gy) will be given to the metastatic lesions. These patients will continue with immunotherapy - Nivolumab and Ipilimumab in accordance with treatment protocol. Approximately one week prior to irradiation a simulation scan will be required. The extent of the low radiation field will depend on the number and location of the metastases, as well as the feasibility and safety of the treatment.

Duration of Therapy

In the absence of treatment delays due to adverse event(s), treatment may continue until one of the following criteria applies:

* Second disease progression
* Intercurrent illness that prevents further administration of treatment
* Unacceptable adverse event(s)
* Patient decides to withdraw from the study
* General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator
* Clinical progression
* Patient non-compliance
* Pregnancy
* Termination of the study by sponsor
* The drug manufacturer can no longer provide the study agent
* In any event medication will not be continued beyond 24 months.

Duration of Follow-Up After removal from study treatment patients will return to the clinic for a short-term FU visit 28 days after the last dose of study treatment.

First long term FU should be performed 100days after the last dose of study drug, and every 90 days thereafter, until death, termination of the study or withdrawal of consent, whichever occurs first. In addition, patients in survival follow-up will be contacted following the data cut-off for the primary analysis and all subsequent survival analyses to provide complete survival data. These contacts should generally occur within 7 days of the data cut off.

* All patients who start the study treatments should be followed up.
* information may be obtained via telephone contact, patient's notes, or public records.
* If the site becomes aware that a patient has died prior to the final analysis, data should be completed at that time.
* Patients who discontinue treatment prior to progression should continue to have RECIST assessments (every 8 weeks from starting study treatment), until confirmed objective disease progression, as defined by RECIST 1.1.

Dose Delay Criteria: Tumor assessments for all subjects should continue as per protocol even if dosing is delayed.

Nivolumab and ipilimumab administration should be delayed for the following:

* Any Grade ≥ 2 non-skin, drug-related adverse event, except for fatigue and laboratory abnormalities
* Any Grade ≥ 3 skin drug-related AE
* Any Grade ≥ 3 drug-related laboratory abnormality with the following exceptions for lymphopenia, AST, ALT, or total bilirubin or asymptomatic amylase or lipase:

  * Grade 3 lymphopenia does not require a dose delay
  * If a subject has a baseline AST, ALT, or total bilirubin that is within normal limits, delay dosing for drug-related Grade ≥ 2 toxicity
  * If a subject has baseline AST, ALT, or total bilirubin within the Grade 1 toxicity range, delay dosing for drug-related Grade ≥ 3 toxicity
  * Any Grade ≥ 3 drug-related amylase or lipase abnormality that is not associated with symptoms or clinical manifestations of pancreatitis does not require dose delay. The Principal Investigator should be consulted for such Grade ≥ 3 amylase or lipase abnormalities.
* Any AE, laboratory abnormality or inter-current illness which, in the judgment of the investigator, warrants delaying the dose of study medication.

Subjects receiving ipilimumab in combination with nivolumab that have drug-related toxicities that meet the criteria for dose delay, should have both drugs (ipilimumab and nivolumab) delayed until retreatment criteria are met. Exceptions apply to the retreatment criteria after dose delay of ipilimumab and nivolumab for Grade ≥ 3 amylase and lipase abnormalities that are not associated with symptoms or clinical manifestations of pancreatitis and that are attributed to ipilimumab alone.

Rescheduling

* Nivolumab may be delayed until the next planned ipilimumab dose if the next ipilimumab dose is scheduled within the next 12 days. This will permit periodic ipilimumab dosing to be synchronized with nivolumab dosing.
* Ipilimumab should be dosed at the specified interval regardless of any delays in intervening nivolumab doses. However, in order to maintain periodic synchronized dosing of ipilimumab and nivolumab, the dosing days of nivolumab and ipilimumab may be adjusted within the permitted +/- 5 day window, as long as consecutive nivolumab doses are given at least 12 days apart. Ipilimumab may be delayed beyond the 5 day window if needed to synchronize with the next nivolumab dose.
* If an ipilimumab dose is delayed beyond 6 weeks from the prior ipilimumab dose, then subsequent ipilimumab doses should rescheduled to maintain the 6 week interval between consecutive ipilimumab doses. Ipilimumab may not be resumed sooner than 6 weeks (+/- 5days) after the prior ipilimumab dose.
* A dose delay of ipilimumab which results in no ipilimumab dosing for > 12 weeks requires ipilimumab discontinuation, with exceptions as noted in study protocol.
* Dose delay of nivolumab which results in treatment interruption of > 6 weeks requires treatment discontinuation, with exceptions as noted

Dose reductions There will be no dose reductions for nivolumab or ipilimumab.

Criteria to Resume Dosing

Subjects may resume treatment with nivolumab and/or ipilimumab when the drug-related AE(s) resolve(s) to Grade ≤ 1 or baseline, with the following exceptions:

* Subjects may resume treatment in the presence of Grade 2 fatigue.
* Subjects who have not experienced a Grade 3 drug-related skin AE may resume treatment in the presence of Grade 2 skin toxicity.
* Subjects with baseline Grade 1 AST/ALT or total bilirubin who require dose delays for reasons other than a 2-grade shift in AST/ALT or total bilirubin may resume treatment in the presence of Grade 2 AST/ALT OR total bilirubin.
* Subjects with combined Grade 2 AST/ALT and total bilirubin values meeting discontinuation parameters should have treatment permanently discontinued.
* Drug-related pulmonary toxicity, diarrhea, or colitis must have resolved to baseline before treatment is resumed.
* For Nivolumab: Subjects with persistent Grade 1 pneumonitis after completion of a steroid taper over at least 1 month may be eligible for retreatment if discussed with and approved by the Principal Investigator.
* Subjects who received systemic corticosteroids for management of any drug-related toxicity must be off corticosteroids or have tapered down to an equivalent dose of prednisone ≤ 10 mg/day.
* Drug-related endocrinopathies adequately controlled with only physiologic hormone replacement may resume treatment after consultation with the Principal Investigator.
* In general, subjects who meet criteria to resume ipilimumab will also have met criteria to resume nivolumab, so it should be feasible to synchronize dosing of both drugs when resuming ipilimumab. In order to facilitate this, the dosing days of nivolumab and ipilimumab may be adjusted within the permitted +/- 5 day window, as long as consecutive nivolumab doses are given at least 12 days apart.
* One exception to note is when ipilimumab and nivolumab doses are delayed due to drug related Grade ≥ 3 amylase or lipase abnormalities not associated with symptoms or clinical manifestations of pancreatitis. If the investigator assesses the amylase or lipase abnormality to be related to ipilimumab and not related to nivolumab, nivolumab may be resumed when the amylase or lipase abnormality resolves to Grade < 3 but ipilimumab may only be resumed when the amylase or lipase abnormality resolves to Grade 1 or baseline. Investigator attribution of this toxicity to the ipilimumab dosing must be clearly noted in the subject's medical chart. The Principal Investigator should be consulted prior to resuming nivolumab in such subjects

Nivolumab Treatment Discontinuation Criteria:

* Any Grade 2 drug-related uveitis or eye pain or blurred vision that does not respond to topical therapy and does not improve to Grade 1 severity within the re-treatment period OR requires systemic treatment.
* Any Grade ≥ 2 drug-related pneumonitis or interstitial lung disease that does not resolve to dose delay and systemic steroids (also see Pulmonary Adverse Event Management Algorithm).
* Any Grade 3 drug-related bronchospasm, hypersensitivity reaction, or infusion reaction, regardless of duration.
* Any Grade 3 non-skin, drug-related adverse event lasting > 7 days, with the following exceptions for uveitis, pneumonitis, bronchospasm, diarrhea, colitis, neurologic toxicity, hypersensitivity reactions, infusion reactions, endocrinopathies, and laboratory abnormalities:

  * Grade 3 drug-related uveitis, pneumonitis, bronchospasm, diarrhea, colitis, neurologic toxicity, hypersensitivity reaction, or infusion reaction of any duration requires discontinuation.
  * Grade 3 drug-related endocrinopathies adequately controlled with only physiologic hormone replacement do not require discontinuation.
  * Grade 3 drug-related laboratory abnormalities do not require treatment discontinuation except:
  * Grade 3 drug-related thrombocytopenia > 7 days or associated with bleeding requires discontinuation.
  * Any drug-related liver function test (LFT) abnormality that meets the following criteria require discontinuation (also see Hepatic Adverse Event Management Algorithm):

    * AST or ALT > 5-10 x ULN for > 2 weeks
    * Total bilirubin > 5 x ULN
    * Concurrent AST or ALT > 3 x ULN and total bilirubin > 2 x ULN
* Any Grade 4 drug-related adverse event or laboratory abnormality, except for the following events, which do not require discontinuation:

  * Grade 4 neutropenia ≤ 7 days
  * Grade 4 lymphopenia or leukopenia
  * Isolated Grade 4 amylase or lipase abnormalities that are not associated with symptoms or clinical manifestations of pancreatitis and decrease to < Grade 4 within 1 week of onset. The Principal Investigator should be consulted for Grade 4 amylase or lipase abnormalities
  * Isolated Grade 4 electrolyte imbalances/abnormalities that are not associated with clinical sequelae and are corrected with supplementation/appropriate management within 72 hours of their onset
  * Grade 4 drug-related endocrinopathy adverse events such as adrenal insufficiency, ACTH deficiency, hyper- or hypothyroidism, or glucose intolerance, which resolve or are adequately controlled with physiologic hormone replacement (corticosteroids, thyroid hormones) or glucose controlling agents, respectively, may not require discontinuation after discussion with and approval from the Principal Investigator.
  * Dosing delays lasting > 6 weeks that occur for non-drug-related reasons may be allowed if approved by the Principal Investigator. Periodic study visits to assess safety and laboratory studies should also continue every 6 weeks or more frequently if clinically indicated during such dosing delays.
* Any adverse event, laboratory abnormality, or intercurrent illness which, in the judgment of the Investigator, presents a substantial clinical risk to the subject with continued ivolumab dosing.

If discontinuation criteria are met for ipilimumab but not for nivolumab, treatment with nivolumab may continue.

Ipilimumab Treatment Discontinuation Criteria:

* Any Grade ≥ 2 drug-related uveitis or eye pain or blurred vision that does not respond to topical therapy and does not improve to Grade 1 severity within 2 weeks OR requires systemic treatment.
* Any Grade ≥3 bronchospasm or other hypersensitivity reaction.
* Any other Grade 3 non-skin, drug-related adverse with the following exceptions for laboratory abnormalities, grade 3 nausea and vomiting, grade 3 neutropenia and thrombocytopenia, and symptomatic endocrinopathies which resolved (with or without hormone substitution).
* Any drug-related liver function test (LFT) abnormality that meets the following criteria require discontinuation:

AST or ALT > 8 x ULN Total bilirubin > 5 x ULN Concurrent AST or ALT > 3 x ULN and total bilirubin > 2 x ULN

* Any Grade 4 drug-related adverse event or laboratory abnormality, except for the following events, which do not require discontinuation:

  * Grade 4 neutropenia ≤ 7 days
  * Grade 4 lymphopenia or leukopenia
  * Isolated Grade 4 amylase or lipase abnormalities which are not associated with symptoms or clinical manifestations of pancreatitis.
  * Isolated Grade 4 electrolyte abnormalities that are not associated with clinical sequelae and are corrected with appropriate management within 72 hours of their onset
  * Grade 4 drug-related endocrinopathy adverse events such as adrenal insufficiency, ACTH deficiency, hyper- or hypothyroidism, or glucose intolerance, which resolve or are adequately controlled with physiologic hormone replacement or glucose controlling agents, respectively, may not require discontinuation after discussion with the Principal Investigator.
* Dosing delays resulting in no ipilimumab dosing for > 12 weeks that occur for non-drug-related reasons may be allowed if approved by the Principal Investigator.
* Any adverse event, laboratory abnormality, or intercurrent illness which, in the judgment of the Investigator, presents a substantial clinical risk to the subject with continued ipilimumab dosing

Treatment Beyond Disease Progression 2

Subjects will be permitted to continue on nivolumab and ipilimumab for treatment beyond initial RECIST v1.1 defined PD as long as they meet the following criteria:

* Investigator-assessed clinical benefit and no rapid disease progression
* Subject is tolerating study treatment
* Stable performance status
* Treatment beyond progression will not delay an imminent intervention to prevent serious complications of disease progression (e.g., CNS metastases) A follow-up scan should be performed within 4 weeks ±5 days of original PD to determine whether there has been a continued progression of disease. Subsequent scans should be performed every 8 weeks until further progression is determined.

Study treatment should be discontinued permanently upon further progression.

ADVERSE EVENTS: LIST AND REPORTING REQUIREMENTS AEs will be graded and recorded throughout the trial and during the follow-up period according to NCI CTCAE Version 5.0. Toxicities will be characterized in terms regarding seriousness, causality, toxicity grading, and action taken with regard to trial treatment.

Identifying the adverse event:

Any inflammatory event, especially those that may respond to steroids, should be considered a possible adverse event. Most such events cannot be identified on physical examination. It should be appreciated that patients may not report these symptoms, or may present to other specialists, who may give inappropriate treatment, e.g potent anti-diarrheal to control a resistant diarrhea. Furthermore, physicians should be aware that some side effects may appear many weeks after treatment initiation.

Early diagnosis and treatment intervention for inflammatory events can help prevent the occurrence of complications, such as GI perforation. Toxicities related to GI (diarrhea and colitis) and skin (rash and pruritus) are the most common inflammatory events reported in studies with ipilimumab.

The combination of both Nivolumab+ipilimumab results in a safety profile with similar types of AEs as either agent alone, but in some cases, with a greater frequency. In general, dose delays and observation are adequate for low-grade AEs. For moderate- and high-grade AEs, immunosuppression with corticosteroids should be utilized. Once the AE has begun to improve, corticosteroids can be tapered over approximately 3 weeks to 6 weeks (depending on the severity of the AE). The management of AEs considered related to any combination treatment is similar to the management of AEs caused by either agent alone and utilizes the same safety management algorithms.

Patients should be assessed for signs and symptoms of enterocolitis, dermatitis, neuropathy, and endocrinopathy; and clinical chemistries (including liver function and thyroid function tests) should be evaluated at baseline and at regular intervals.

Overview of management of adverse event Aside from very mild side effects, the first step should be to hold all study immunotherapies. Early intervention with steroids is to be considered in the majority of cases, followed possibly by re-starting the study therapeutic agents.

During evaluation of a suspected immune-mediated AE, all efforts should be made to rule out neoplastic, infectious, metabolic, toxic, or other etiologic causes. Serological, immunological, imaging, and occasionally biopsy with histology (e.g., biopsy-proven lymphocytic) data may be used to support the diagnosis of an immune-mediated toxicity or support an alternative cause of the AE.

In general, for severe immune-mediated AEs, nivolumab and/or ipilimumab should be permanently discontinued, and systematic high-dose corticosteroid therapy should be initiated. For moderate immune-mediated AEs, ipilimumab should be held or delayed, and moderate-dose corticosteroids should be considered. Upon improvement, corticosteroids should be tapered gradually over at least 1 month.

The causal relationship to study drug is determined by a physician and should be used to assess all adverse events (AE).

Definition of Serious Adverse Event Serious events include, but are not limited to, intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization.) Potential drug induced liver injury (DILI) is also considered an important medical event.

Suspected transmission of an infectious agent via the study drug is an SAE. Although pregnancy, overdose, cancer, and potential drug induced liver injury (DILI) are not always serious by regulatory definition, these events must be handled as SAEs. Any component of a study endpoint that is considered related to study therapy should be reported as SAE.

NOTE: The following hospitalizations are not considered SAEs:

* a visit to the emergency room or other hospital department < 24 hours
* elective surgery, planned prior to signing consent
* routine health assessment requiring admission for baseline/trending of health status (eg, routine colonoscopy).
* Medical/surgical admission other than to remedy ill health and planned prior to entry into the study.
* Admission encountered for another life circumstance that carries no bearing on health status and requires no medical/surgical intervention.
* Admission for administration of anticancer therapy in the absence of any other SAEs (applies to oncology protocols)

Serious Adverse Event Collection and Reporting All SAEs must be collected that occur during the screening period and within 100 days of the last dose of study drug. Subjects, who are randomized and never treated with study drug, must have SAEs collected for 30 days from the date of randomization. If applicable, SAEs that relate to any later protocol-specified procedure (eg, a follow-up skin biopsy) must be collected.

The investigator should report any SAE that occurs after these time periods and that is believed to be related to study drug or protocol-specified procedure.

An SAE report should be completed for any event where doubt exists regarding its seriousness.

If the investigator believes that an SAE is potentially related to the conditions of the study (such as withdrawal of previous therapy or a complication of a study procedure), the relationship should be specified.

SAEs, whether related or not related to study drug, and pregnancies must be reported to BMS (or designee) within 24 hours of awareness of event. SAEs must be recorded on the SAE Report Form; pregnancies on a Pregnancy Surveillance Form. Paper forms are to be transmitted via email or confirmed facsimile (fax). In addition, the local IRB will be informed per local regulations.

If only limited information is initially available, follow-up reports are required. (Note: Follow-up SAE reports should include the same investigator term(s) initially reported.) If an ongoing SAE changes in its intensity or relationship to study drug or if new information becomes available, a follow-up SAE report should be sent within 24 hours to BMS (or designee) using the same procedure.

All SAEs should be followed to resolution or stabilization. The Investigator will request from BMS the SAE reconciliation report and include the BMS protocol number every 3 months and prior to data base lock or final data summary.

Nonserious Adverse Event Collection and Reporting The collection of non-serious AE information should begin following the subject's written consent to participate in the study And should be followed to resolution or stabilization of the adverse event to grade 1, or reported as SAEs if they become serious. Follow-up is also required for nonserious AEs that cause interruption or discontinuation of study drug and for those present at the end of study treatment as appropriate. All AEs must be recorded on the CRF.

All nonserious adverse events are to be collected continuously during the treatment period and for a minimum of 28 days following the last dose of study treatment.

Pregnancy Investigator must immediately notify BMS of Pregnancy event and complete and forward a Pregnancy Surveillance Form within 24 hours of awareness of the event and in accordance with SAE reporting procedures.

In the rare event that the benefit of continuing study drug is thought to outweigh the risk, the pregnant subject may continue study drug after a thorough discussion, if allowed by local regulations.

Protocol-required procedures for study discontinuation and follow-up must be performed on the subject unless contraindicated by pregnancy (eg, x-ray studies). Other appropriate pregnancy follow-up procedures should be considered if indicated.

Follow-up information regarding the course of the pregnancy, including perinatal and neonatal outcome and, where applicable, offspring information must be reported on the Pregnancy Surveillance Form.

Men receiving nivolumab and who are sexually active with women of childbearing potential will be instructed to adhere to contraception for a period of 7 months after the last dose of nivolumab.

In order to collect any pregnancy surveillance information from the female partner, the female partner must sign an informed consent form for disclosure of this information. Information on this pregnancy will be collected on the Pregnancy Surveillance Form and reported to BMS.

Overdose An overdose is defined as the accidental or intentional administration of any dose of a product that is considered both excessive and medically important. All occurrences of overdose must be reported as SAEs.

Potential Drug Induced Liver Injury (DILI) All occurrences of potential DILIs, meeting the defined criteria, must be reported as SAEs .

Potential DILI is defined as: ALT or AST elevation > 3 times upper limit of normal (ULN) AND Total bilirubin > 2 times ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase), AND No other immediately causes of AT elevation and hyperbilirubinemia.

A hepatic AE management algorithm has been established (and is indicated in the protocol).

CORRELATIVE STUDIES During IO therapy Blood, Stool and Saliva samples for correlative study will be taken cycle 1 Day 1 of and every 8 weeks thereafter. Biopsies of the disease lesion will be obtained prior to start of treatment and at 8 weeks. Specific permission will therefore be included in the consent form. Local regulations for tissue banking and storage will be followed.

Fresh biopsy specimens from disease lesion during screening (preferably, at site of SBRT) and at 8 weeks imaging assessment are mandatory. Optional tissue biopsy will be requested at progression. (For patients that have stopped treatment for other reasons than PD, tissue biopsy will be requested at the time of PD.

In addition, Tissue samples will be submitted from existing archived biopsy (diagnostic specimen), if available.

STATISTICAL CONSIDERATIONS

Study populations will include safety and efficacy:

* Safety Population will include all subjects who receive at least 1 dose of ipilimumab, nivolumab.
* Efficacy population will include all subjects in the Safety Population with at least 1 recorded post-baseline disease assessment Statistical methods will be primarily descriptive in nature. Categorical variables will be summarized using numbers and percentages. Continuous variables will be summarized by total number (n), mean, standard deviation, median, and range (minimum and maximum).

Event rates will be summarized, and Kaplan-Meier estimates for PFS and OS may also be provided where sample size is adequate.

Safety data, including vital signs, laboratory test results, physical examinations, and adverse events (AEs), will be summarized by dose and assessment time points, as appropriate. Change from baseline will be included in summary tables for laboratory, and vital sign parameters.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent and be between the ages of 18 and up.
* Metastatic histology proven adenocarcinoma of the pancreas. If patient has primary resected tumor, tumor recurrence needs to >12 months after last adjuvant chemotherapy.
* ECOG performance status 0-1.
* Life expectancy of >= 3 months.
* If female and of child-bearing potential, have a negative serum pregnancy test during screening.
* Agree to use of a barrier method of contraception if sexually active (both men and women) from the time of administration of the first treatment and for at least 5 months after treatment.
* Have PT - INR < 1.5, WBC > 2000/μL absolute neutrophil count (ANC) > 1500 x 103 cells/ μL, platelets ≥ 100,000/ μL, and hemoglobin >= 9 mg/dL Serum creatinine < 1.5 x ULN, unless creatinine clearance ≥ 40 mL/min (measured or calculated using the Cockroft-Gault formula) AST/ALT: < 3.0 x ULN Total bilirubin < 1.5 x ULN (except participants with Gilbert Syndrome who must have a total bilirubin level of < 3.0x ULN).
* A disease lesion, including primary pancreas lung/liver/peritoneal/bone /lynph nodes, that is suitable for SBRT as deemed by the investigator.
* Screening procedures completed within 4 weeks of starting treatment.
* Availability of at least 1 measurable lesion not previously irradiated that is not planned to be irradiated with SBRT during the study and measurable as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Patient received minimum of 4 cycles of first-line chemotherapy of induction chemotherapy per investigator's decision without progression.
* Adjuvant treatment is allowed if ≥ 12 months has passed since last adjuvant treatment.
* Fresh biopsy specimens are required unless biopsy deemed unsafe by investigator.

Exclusion Criteria:

* Clinically significant pancreatitis within 8 weeks of treatment.
* Pregnant and breastfeeding women are excluded. Women of child-bearing potential who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period and for up to 5 months after the study are excluded.
* A medical condition or any intercurrent medical illness or other medical condition that would in the judgment of the investigator compromise patient safety or the objectives of the study.
* Have participated in any therapeutic research study within the last 4 weeks.
* Known medical condition that predisposes to radiation toxicity (e.g. scleroderma)
* Has a known MSI-H phenotype or a known MMR deficiency.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with type I diabetes mellitus, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll. Subjects that require intermittent use of bronchodilators or local steroids, e.g., inhaled or topical steroids, at a dose of less than the equivalent of 10mg prednisone daily, would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial (chronic pain management medications should not exclude study participation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective tumor response rate1 (ORR1) in study patients, assessed by RECIST v1.1 | From first dose of SBRT until first progression, approximately 36 months.
  Proportion of subjects showing best overall response of complete response (CR) or partial response (PR)
Objective tumor response rate 2 (ORR2) after first progression, assessed by RECIST v1.1 | From the date of low dose radiation until second progression, approximately 36 months
  Proportion of subjects with best overall response of CR or PR, in progressors who continue to receive low dose radiation and re-challenge nivolumab and ipilimumab

SECONDARY OUTCOMES:
Progression free survival 1 (PFS 1) in stage 4 PDAC, assessed by RECIST 1.1 | From first dose of SBRT until first progression, approximately 36 months
  Duration of time from first dose of SBRT until confirmed objective disease progression or death (or date of last documentation of being alive).
Objective tumor progression free survival 2 (PFS 2) in progressors, assessed by RECIST v1.1 | From the date of low dose radiation until second progression, approximately 36 months
  Duration of time until 2nd confirmed objective disease progression or death (or last documentation of being alive).
Median Overall survival (OS) | From documented metastatic disease until death (or date of last documentation of being alive), approximately 36 months
  Duration of time from diagnosis until death (or date of last documentation of being alive). Survival data may be obtained via contact with the patient, patient's family, or through a review of the patient's notes, or through the use of public records.
Incidence of Treatment-Emergent Adverse Events, as assessed by CTCAE version 5.0 | From day of subject's written consent until study termination, approximately 36 months
  Any new condition or change from baseline will be included in summary tables.

OTHER OUTCOMES:
Assessment of disease biomarkers as a surrogates or predictors to response following administration of SBRT and immunotherapy: Exploratory | 5 years
  Blood and tumor samples will be analyzed for various biomarkers. Initial biomarkers to be tested include proteins such as PDL-1, functional DNA repair assays, stromal elements, immune cells ratio, DNA and RNA next generation sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Talia Golan, Prof., Principal Investigator — Shaba Medical Center
Locations (1):
- Sheba Medical Centre, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Demaria S, Golden EB, Formenti SC. Role of Local Radiation Therapy in Cancer Immunotherapy. JAMA Oncol. 2015 Dec;1(9):1325-32. doi: 10.1001/jamaoncol.2015.2756. PMID 26270858
- [Background] Menon H, Chen D, Ramapriyan R, Verma V, Barsoumian HB, Cushman TR, Younes AI, Cortez MA, Erasmus JJ, de Groot P, Carter BW, Hong DS, Glitza IC, Ferrarotto R, Altan M, Diab A, Chun SG, Heymach JV, Tang C, Nguyen QN, Welsh JW. Influence of low-dose radiation on abscopal responses in patients receiving high-dose radiation and immunotherapy. J Immunother Cancer. 2019 Sep 4;7(1):237. doi: 10.1186/s40425-019-0718-6. PMID 31484556
- [Background] Wolchok JD, Kluger H, Callahan MK, Postow MA, Rizvi NA, Lesokhin AM, Segal NH, Ariyan CE, Gordon RA, Reed K, Burke MM, Caldwell A, Kronenberg SA, Agunwamba BU, Zhang X, Lowy I, Inzunza HD, Feely W, Horak CE, Hong Q, Korman AJ, Wigginton JM, Gupta A, Sznol M. Nivolumab plus ipilimumab in advanced melanoma. N Engl J Med. 2013 Jul 11;369(2):122-33. doi: 10.1056/NEJMoa1302369. Epub 2013 Jun 2. PMID 23724867
- [Background] Milas L, Mason KA, Ariga H, Hunter N, Neal R, Valdecanas D, Krieg AM, Whisnant JK. CpG oligodeoxynucleotide enhances tumor response to radiation. Cancer Res. 2004 Aug 1;64(15):5074-7. doi: 10.1158/0008-5472.CAN-04-0926. PMID 15289307
- [Background] Formenti SC, Demaria S. Combining radiotherapy and cancer immunotherapy: a paradigm shift. J Natl Cancer Inst. 2013 Feb 20;105(4):256-65. doi: 10.1093/jnci/djs629. Epub 2013 Jan 4. PMID 23291374